CLINICAL TRIAL: NCT06393907
Title: A Randomized Trial of Hemostatic Forceps Versus Bipolar Electrocautery Probes for High-Risk Bleeding Gastroduodenal Ulcers
Brief Title: Hemostatic Forceps vs. Bipolar Electrocautery Probes for High-Risk Bleeding Gastroduodenal Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Uayporn, Assistant professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si 223/2024
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Gastroduodenal Ulcer
Keywords: Hemostatic Forceps; Bipolar Electrocautery Probes; Gastroduodenal Ulcer; Rebleeding; Hemostasis; Peptic ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Intervention Model Description: Hemostatic Forceps versus Bipolar Electrocautery Probes
Who Masked: Participant
Masking Description: The participants will be randomized for each intervention using sequentially numbered, opaque sealed envelopes after recruitment in the study. The care provider who uses the devices cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hemostatic forceps (Experimental): Hemostatic forceps will be used for control bleeding with electrocautery unit setting: 80 W, effect 4, soft coagulation mode for 1-2 seconds.
  Interventions: Device: Hemostatic Forceps
- Bipolar electrocautery probes (Active Comparator): Bipolar electrocautery probes will be used for control bleeding with electrocautery unit setting: effect 2, soft coagulation bipolar mode for 8-10 seconds.
  Interventions: Device: Bipolar Electrocautery Probes

INTERVENTIONS:
Device: Hemostatic Forceps — The experimental device will be used for control bleeding in high risk gastroduodenal ulcers.
  Other Names: Coagrasper (Olympus, Tokyo, Japan)
  Arms: Hemostatic forceps
Device: Bipolar Electrocautery Probes — The active comparator devices will be used for control bleeding in high risk gastroduodenal ulcers.
  Other Names: Gold probe (Boston Scientific, Massachusetts, USA)
  Arms: Bipolar electrocautery probes

SUMMARY:
A randomized controlled trial to evaluate the efficacy of hemostatic forceps and bipolar electrocautery probes in patient with high risk bleeding gastroduodenal ulcers.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial to evaluate the efficacy of hemostatic forceps and bipolar electrocautery probes in patients with high-risk bleeding gastroduodenal ulcers. The primary outcome is comparing the hemostatic rates of the devices. Secondary outcomes are rebleeding rate at 7 and 30 days after index intervention, survival rate after intervention, procedure time for achieving hemostasis, number of units of infused blood, duration of hospitalization, and complications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient with upper gastrointestinal hemorrhage age ≥ 18 years old
2. The patient with gastroduodenal ulcer with indication for hemostatic intervention including 2.1 Forrest classification 1a (Active spurting) 2.2 Forrest classification 1b (Active oozing) 2.3 Forrest classification 2a (Non-bleeding visible vessel; NBVV) 2.4 Forrest classification 2b (Adherent clot) with lesion underneath clot which need hemostatic intervention including active spurting, active oozing or non-bleeding visible vessel

Exclusion Criteria:

1. Uncorrectable hemostasis laboratory including serum platelet < 50000 /mm3 or International Normalized Ratio (INR) >1.5
2. Bleeding from cancerous gastroduodenal ulcer
3. The patient with history of gastric surgery
4. The patient with history of bleeding gastroduodenal ulcer within 30 days prior to enrollment
5. The patient with history of proton pump inhibitor allergy
6. Pregnant
7. The patient deny to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Comparing hemostatic rate between hemostatic forceps and bipolar electrocautery probes | During esophagogastroduodenoscopy
  When the bleeding stopped for at least 2 minutes, it is defined as successful hemostasis.

SECONDARY OUTCOMES:
Rebleeding rate at 7 days and 30 days after index intervention | 30 days
  After primary hemostasis, patients will be follow up at 7 and 30 days for evidence of rebleeding.
Survival rate after intervention | 30 days
  Patients who live longer than 30 days after hemostasis will be counted for survival rate.
Procedure time for achieving hemostasis | During esophagogastroduodenoscopy
  Procedure time will be counted from the time of device insertion to the time of achieving hemostasis.
Number of units of infused blood | 30 days
  Number of red cell units which are transfused to the patients.
Duration of hospitalization | 30 days
  The length of hospital stay.
Complications of hemostatic interventions | 30 days
  Complications related to intervention include perforation, infection, and organ failure

CONTACTS AND LOCATIONS:
Overall Officials: Uayporn Kaosombatwattana, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of internal medicine siriraj hospital, Mahidol university, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Background] Charatcharoenwitthaya P, Pausawasdi N, Laosanguaneak N, Bubthamala J, Tanwandee T, Leelakusolvong S. Characteristics and outcomes of acute upper gastrointestinal bleeding after therapeutic endoscopy in the elderly. World J Gastroenterol. 2011 Aug 28;17(32):3724-32. doi: 10.3748/wjg.v17.i32.3724. PMID 21990954
- [Background] Forrest JA, Finlayson ND, Shearman DJ. Endoscopy in gastrointestinal bleeding. Lancet. 1974 Aug 17;2(7877):394-7. doi: 10.1016/s0140-6736(74)91770-x. No abstract available. PMID 4136718
- [Background] ASGE technology committee; Parsi MA, Schulman AR, Aslanian HR, Bhutani MS, Krishnan K, Lichtenstein DR, Melson J, Navaneethan U, Pannala R, Sethi A, Trikudanathan G, Trindade AJ, Watson RR, Maple JT; ASGE Technology Committee Chair. Devices for endoscopic hemostasis of nonvariceal GI bleeding (with videos). VideoGIE. 2019 Jun 27;4(7):285-299. doi: 10.1016/j.vgie.2019.02.004. eCollection 2019 Jul. PMID 31334417
- [Background] Asge Technology Committee; Conway JD, Adler DG, Diehl DL, Farraye FA, Kantsevoy SV, Kaul V, Kethu SR, Kwon RS, Mamula P, Rodriguez SA, Tierney WM. Endoscopic hemostatic devices. Gastrointest Endosc. 2009 May;69(6):987-96. doi: 10.1016/j.gie.2008.12.251. No abstract available. PMID 19410037
- [Background] Arima S, Sakata Y, Ogata S, Tominaga N, Tsuruoka N, Mannen K, Shiraishi R, Shimoda R, Tsunada S, Sakata H, Iwakiri R, Fujimoto K. Evaluation of hemostasis with soft coagulation using endoscopic hemostatic forceps in comparison with metallic hemoclips for bleeding gastric ulcers: a prospective, randomized trial. J Gastroenterol. 2010 May;45(5):501-5. doi: 10.1007/s00535-009-0186-8. Epub 2009 Dec 25. PMID 20033825
- [Background] Kim JW, Jang JY, Lee CK, Shim JJ, Chang YW. Comparison of hemostatic forceps with soft coagulation versus argon plasma coagulation for bleeding peptic ulcer--a randomized trial. Endoscopy. 2015 Aug;47(8):680-7. doi: 10.1055/s-0034-1391565. Epub 2015 Mar 2. PMID 25730283
- [Background] Nunoue T, Takenaka R, Hori K, Okazaki N, Hamada K, Baba Y, Yamasaki Y, Kono Y, Seki H, Inokuchi T, Takemoto K, Taira A, Tsugeno H, Fujiki S, Kawahara Y, Okada H. A Randomized Trial of Monopolar Soft-mode Coagulation Versus Heater Probe Thermocoagulation for Peptic Ulcer Bleeding. J Clin Gastroenterol. 2015 Jul;49(6):472-6. doi: 10.1097/MCG.0000000000000190. PMID 25083773
- [Background] Toka B, Eminler AT, Karacaer C, Uslan MI, Koksal AS, Parlak E. Comparison of monopolar hemostatic forceps with soft coagulation versus hemoclip for peptic ulcer bleeding: a randomized trial (with video). Gastrointest Endosc. 2019 Apr;89(4):792-802. doi: 10.1016/j.gie.2018.10.011. Epub 2018 Oct 17. PMID 30342026
- [Background] Bianco MA, Rotondano G, Marmo R, Piscopo R, Orsini L, Cipolletta L. Combined epinephrine and bipolar probe coagulation vs. bipolar probe coagulation alone for bleeding peptic ulcer: a randomized, controlled trial. Gastrointest Endosc. 2004 Dec;60(6):910-5. doi: 10.1016/s0016-5107(04)02232-1. PMID 15605005
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Veitch AM, Radaelli F, Alikhan R, Dumonceau JM, Eaton D, Jerrome J, Lester W, Nylander D, Thoufeeq M, Vanbiervliet G, Wilkinson JR, Van Hooft JE. Endoscopy in patients on antiplatelet or anticoagulant therapy: British Society of Gastroenterology (BSG) and European Society of Gastrointestinal Endoscopy (ESGE) guideline update. Gut. 2021 Sep;70(9):1611-1628. doi: 10.1136/gutjnl-2021-325184. PMID 34362780